CLINICAL TRIAL: NCT04043559
Title: Small Cortical Cerebellar Infarctions Are Associated With Patent Foramen Ovale in Young Cryptogenic Stroke Patients
Brief Title: Cortical Cerebellar Infarctions Associated With Patent Foramen Ovale in Young Stroke Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2019/DR-01
Record Dates: First submitted 2019-07-25; First posted 2019-08-02 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2021-09

CONDITIONS: Brain Infarction
MeSH Terms: conditions — Brain Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with an acute symptomatic infarction
  Interventions: Other: MRI scanner; Other: Contrast transoesophageal echocardiography
- controls with cryptogenic stroke
  Interventions: Other: MRI scanner; Other: Contrast transoesophageal echocardiography

INTERVENTIONS:
Other: MRI scanner — MRI was performed with a 1.5T magnet (Ingenia, Philips, The Netherlands; diffusion-weighted imaging b-values = 0 and 1,000 s/mm2, TR 4,280 ms, and TE 97 ms). In case of technical problems with the 1.5T MRI scanner, a 3T magnet (Skyra, Siemens, Erlangen, Germany) was used. MRI was analyzed by an experienced rater (DR), blinded to clinical data and MRI sequences other than diffusion-weighted imaging.
Other: Contrast transoesophageal echocardiography — Contrast transoesophageal echocardiography (including Valsalva manoeuvre)

SUMMARY:
The investigator retrospectively analyzed consecutive young (<60 years) cryptogenic stroke patients with Patient Foramen Ovale (PFO) recruited between January 2016 and May 2019 in our center, and compared these patients with sex- and age-matched controls with cryptogenic stroke without PFO. Analyzed baseline characteristics: sex, age, cardiovascular risk factors, history of stroke, and cortical/subcortical localization, arterial territory, number of lesions, and lesion size of the acute symptomatic infarction, together with the ROPE score. The presence and the number of acute and chronic SCCI lesions were assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients : young (<60 years) adult patients,
* Patient recruited and registered in our stroke database between January 2016 and May 2016 of our center (Nîmes University Hospital, France),
* Patients presenting with an acute symptomatic infarction (confirmed by diffusion-weighted MRI) of unknown origin
* Controls : age-matched controls with cryptogenic stroke without PFO

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Consecutive young (<60 years) cryptogenic stroke patients with PFO recruited between January 2016 and May 2019 in our center, and compared these patients with sex- and age-matched controls with cryptogenic stroke without PFO.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
number of infarction lesions | day 1
  Number (increase)
infarction location | day 1
  anterior, posterior, or mixed anterior-posterior circulation and the cortical/subcortical/corticosubcortical location of infarction
size of subcortical lesion | day 1
  < or >15mm
presence of multiterritorial infarction | day 1
  mixed anterior-posterior circulation or bilateral anterior circulation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nîmes, Nîmes, France

REFERENCES:
- [Result] Renard D, Ion I, Ricci JE, Mura T, Thouvenot E, Wacongne A. Chronic Small Cortical Cerebellar Infarctions on MRI are Associated with Patent Foramen Ovale in Young Cryptogenic Stroke. Cerebrovasc Dis. 2020;49(1):105-109. doi: 10.1159/000505959. Epub 2020 Feb 14. PMID 32062661